CLINICAL TRIAL: NCT03565003
Title: A Phase 1/2a, Multi-Center, Dose Escalation/Dose Expansion, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Evidence of Antitumor Activity of JAB-3068 in Adult Patients With Advanced Solid Tumors
Brief Title: A First-in-Human Study of JAB-3068 (SHP2 Inhibitor) in Adult Patients With Advanced Solid Tumors in China
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jacobio Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JAB-3068-02
Record Dates: First submitted 2018-05-29; First posted 2018-06-21 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2022-03

CONDITIONS: Non-small Cell Lung Cancer; Head and Neck Cancer; Esophageal Cancer; Other Metastatic Solid Tumors
Keywords: JAB-3068; SHP2; PTPN11; ESCC; NSCLC; HNSCC; Colorectal cancer (CRC); EGFR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms; Esophageal Neoplasms; Noonan Syndrome; Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JAB-3068 (SHP2 inhibitor) (Experimental): JAB-3068 will be administered orally in the morning following a fast of approximately 6 hours before on PK collection. Patients will continue to fast for approximately 2 hours after the administration of JAB-3068. On non-PK days patients will fast approximately 2 hours before JAB-3068 and continue to fast for approximately 2 hours afterwards.
  Interventions: Drug: JAB-3068

INTERVENTIONS:
Drug: JAB-3068 — 25 mg,100 mg

SUMMARY:
This is a Phase 1/2a, open-label, multi-center study of JAB-3068 in Patients with advanced solid tumors.This study has two phases: dose escalation phase and dose expansion phase.

DETAILED DESCRIPTION:
Dose escalation study phase is designed to determine the maximum tolerated dose (MTD) according to a 3+3 design and recommended phase II dose (RP2D) and to characterize the safety, tolerability, and pharmacokinetics (PK) profile of JAB-3068. Other dose regimens may be explored based on the analysis of emerging PK and safety data. at this study phase, JAB-3068 dministered orally once daily (QD) or twice daily (BID) or once every other day (QOD) in 28-day treatment cycles to adult patients with advanced solid tumors,

Dose expansion study phase is designed to evaluate the antitumor activity(ORR and DOR) of JAB-3068 in patients with NSCLC, ESCC and HNSCC.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study-related procedure being performed;
2. Age 18 years or older;
3. Dose escalation(phase I): Patients with histologically or cytologically confirmed, advanced solid tumors (including lymphoma) which have progressed from standard therapy or for whom no standard therapy exists; Dose expansion(phase IIa ): Patients with histologically or cytologically confirmed, advanced NSCLC, ESCC, HNSCC which have progressed from standard therapy;
4. Patients with life expectancy ≥3 months;
5. Dose expansion(phase IIa ): patients have available archival tissue can be provided or willing to perform biopsy to provide fresh tumor tissue.
6. Patients with other solid tumors must have at least one measurable lesion as defined by RECIST v1.1;Patients with Lymphomas must have at least one measurable lesion as defined by IWG 2007 criteria;
7. Eastern Cooperative Oncology Group performance score 0 or 1;
8. Patients who have sufficient baseline organ function.

Exclusion Criteria:

1. Patients with life-threatening autoimmune disease or with autoimmune disorder and who are on long-term steroid treatment;
2. History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO;
3. Lymphoma with brain metastasis; Other solid tumors:Known malignant central nervous system (CNS) disease other than neurologically stable, treated brain metastases;
4. Active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV)
5. Patients who have any severe and/or uncontrolled medical conditions or other conditions that, in the opinion of the Investigator and Sponsor, could affect the patient's participation in the study
6. Patients who have impaired cardiac function or clinically significant cardiac diseases
7. Use of anti-cancer treatment drug ≤21 days prior to the first dose of JAB-3068.
8. Use of an investigational drug during the past 30 days prior to the first dose of JAB-3068.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities | At the end of Cycle 1 (each cycle is 28 days)
  Number of participants with dose limiting toxicities (DLTs) in the dose escalation phase. A DLT is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first treatment cycle with JAB-3068.
Objective response rate | Approximately 2 years
  ORR is defined as the proportion of participants with complete response or partial. the ORR of JAB-3068 in patients with ESCC, NSCLC and HNSCC will be evaluated separately in dose expansion
Duration of response | Approximately 2 years
  DOR is defined as the time from the participant's initial objective response (CR or PR) to study drug therapy, to disease progression or death due to any cause, whichever occurs first. The DOR of JAB-3068 in patients with ESCC, NSCLC and HNSCC will be evaluated separately in dose expansion

SECONDARY OUTCOMES:
Number of participants with adverse events | Approximately 2 years
  All patients participating in this study will be assessed for incidence and severity of adverse events (AEs) and serious AEs, including changes in laboratory values, vital signs, electrocardiograms, cardiac imaging and ophthalmological assessments
Area under the curve | Approximately 2 years
  Area under the plasma concentration time curve of JAB-3068
Cmax | Approximately 2 years
  Highest observed plasma concentration of JAB-3068
Tmax | Approximately 2 years
  Time of highest observed plasma concentration of JAB-3068
T1/2 | Approximately 2 years
  Half life of JAB-3068
Objective response rate | Approximately 2 years
  ORR is defined as the proportion of participants with complete response or partial response (CR+PR) in dose escalation.
Duration of response | Approximately 2 years
  DOR is defined as the time from the participant's initial objective response (CR or PR) to study drug therapy, to disease progression or death due to any cause, whichever occurs first in dose escalation.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (4):
- China (4):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chinese PLA Central Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No